CLINICAL TRIAL: NCT05391152
Title: Comparison Between Robotic-Arm Assisted Modified Kinematic Alignment Total Knee Replacement And Traditional Manual Alignment Total Knee Replacement：A Prospective Multicenter, Double-Blind Study
Brief Title: Comparison Between Robotic-arm Assisted Total Knee Replacement and Traditional Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202203
Record Dates: First submitted 2022-05-22; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Knee
Keywords: robotic-arm assisted; total knee replacement; kinematic alignment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic-arm assisted modified kinematic alignment total knee replacement (Experimental): The patients in this group receive robotic-arm assisted total knee replacement. And these patients achieve modified kinematic alignment.
  Interventions: Device: robotic assisted total knee replacement
- traditional manual total knee replacement (Active Comparator): The patients in this group receive traditional manual total knee replacement. And these patients achieve traditional alignment.
  Interventions: Device: traditional total knee replacement

INTERVENTIONS:
Device: robotic assisted total knee replacement — the study group used robotic-arm assisted total knee replacement.
  Arms: robotic-arm assisted modified kinematic alignment total knee replacement
Device: traditional total knee replacement — the control group used traditional total knee replacement
  Arms: traditional manual total knee replacement

SUMMARY:
This is a multicenter, prospective, and case-control study. Five joint centers and 100 participants will be included. The study group used robotic-assisted modified kinematic alignment total knee replacement, and the control study used traditional alignment manual total knee replacement. The knee society score (KSS), Hip-knee-ankle(HKA) angle, mechanical lateral distal femoral angle(mLDFA), mechanical medial proximal tibial angle(mMPTA), sagittal femoral component angle(SFCA), range of motion(ROM), WOMAC score, SF-36, Visual Analogue Scale(VAS score), surgical time, blood loss, and complications are evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 years and 85 years
* primary total knee replacement

Exclusion Criteria:

* obvious bone defect
* infection
* BMI>>35kg/m2
* severe osteoporosis
* mental disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
KSS score | 3 months
  Keen Society Score

SECONDARY OUTCOMES:
HKA angle | 3 months
  hip-knee-ankle angle
mLDFA | 3 months
  mechanical lateral distal femoral angle
mMPTA | 3 months
  mechanical medial proximal tibial angle
SFCA | 3 months
  sagittal femoral component angle
knee ROM | 3 months
  knee range of motion
blood loss | intraoperative
  the intraoperative blood loss
surgical duration | intraoperative
  the duration of the operation
complication | 3 months
  complications after the surgery